CLINICAL TRIAL: NCT06997211
Title: The Effect of the Emotional Freedom Technique Applied to Mothers With Premature Babies in the Intensive Care Unit on Fatigue, Anxiety, and Mother-Baby Bonding
Brief Title: Fatigue, Anxiety, and Mother-Baby Bonding and Emotional Freedom Technique
Acronym: EFT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Merve Meşedüzü, LECTURER, Bezmialem Vakif University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: E-54022451-050.04-171619; MMeseduzu (Other: BezmialemVU)
Record Dates: First submitted 2025-03-03; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Puerperium; EFTs
Keywords: EFT; PRETERM INFANT; ANXIETY; MOTHER-BABY BONDING; FATIGUE; PUERPERIUM
MeSH Terms: conditions — Premature Birth; Anxiety Disorders; Fatigue | interventions — Postpartum Period

STUDY DESIGN:
Intervention Model Description: 1. EFT Procedure Sequence:
  • The first meeting will be conducted within the first 24 hours after the admission of mothers who meet the inclusion criteria for our study in the NICU.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERİMENTAL: EFT GROUP (Experimental): Steps for the Intervention Group:
  Pre-Intervention:
  * Participants in the intervention group will be informed about EFT, and after explaining the aim and method of the study, their consent will be obtained using the Volunteer Consent Form.
  * They will complete the State-Trait Anxiety Inventory (STAI), and those who score 40 or higher will be included in the study.
  * Afterward, information will be provided about EFT, including how the procedure will be performed and how tapping will be done. Following a discussion planned to last approximately 20 minutes, the EFT session will begin.
  * Prior to the intervention, women will be asked to fill out the Descriptive Information Form, State-Trait Anxiety Inventory (STAI-I), Visual Similarity Scale for Fatigue (YİGBS), and Mother-Infant Bonding Scale (MIBS) forms.
    1. EFT Procedure Sequence:
  * The first meeting will be conducted within the first 24 hours after the admission of mothers who meet the inclusion criteria for our study in the NICU.
  * T
  Interventions: Behavioral: EFT
- CONTROL GROUP (No Intervention): Control Group Application Steps:
  Control Group 1st Meeting (Pre-test):
  The mothers in the control group, who have premature babies in the neonatal intensive care unit, will be informed about the study. After explaining the purpose and method of the study, their consent will be obtained through the Volunteer Consent Form.
  The women will complete the forms, and those with a score of 40 or above will be included in the study.
  The women in the control group will be asked to complete the Descriptive Information Form, State-Trait Anxiety Inventory (STAI I-II), Visual Similarity Scale for Fatigue (YİGBS), and Mother-Infant Bonding Scale (MIBS) forms.
  No intervention will be provided for the mothers in the control group, but the institution's neonatal intensive care services will be available to them.
  Control Group 2nd Meeting:
  One week after the first meeting, the State-Trait Anxiety Inventory (STAI I-II), Visual Similarity Scale for Fatigue (YİGBS), and Mother-Infant Bonding Scale (MIBS) fo

INTERVENTIONS:
Behavioral: EFT — The EFT session will be conducted mutually with the practitioner. The average duration of the session is planned to be 40-45 minutes.
  Other Names: EFT AND PUERPERIUM
  Arms: EXPERİMENTAL: EFT GROUP

SUMMARY:
Fatigue, Anxiety, and Mother-Baby Bonding and Emotional Freedom Technique

DETAILED DESCRIPTION:
Type of research: This study is a randomized controlled experimental study designed according to the Consolidated Standards of Reporting Trials (CONSORT) guideline.

Place of the research: Bezmialem Vakıf University Central Hospital Neonatal Intensive Care Unit and Obstetrics and Gynecology Service, Bezmialem Vakıf University Dragos Hospital Neonatal Intensive Care Unit and gynecology service.

Population of the Research: The population of the research consists of mothers of premature newborns who were hospitalized in Bezmialem Vakıf University Central Hospital Neonatal Intensive Care Unit and Bezmialem Vakıf University Dragos Hospital Newborn Intensive Care Unit on the study dates.

Research Sample: Power analysis was conducted to determine the number of people to be included in the research. The power of the test was calculated with the G*Power 3.1 program. the effect size regarding state anxiety change was calculated as 0.866. In order to exceed the 99% value in determining the power of the study; At a significance level of 5% and an effect size of 0.866, 54 people, 27 people in the groups, need to be reached (df=26; t=2.056). In the research, it was aimed to reach a total of 64 people, 32 people in the groups, considering the high power of the test and the losses.

Analysis of Data: It was planned to use SPSS (Statistical Package for Social Sciences) for Windows 22.0 program for the statistics of the data obtained in the research. Number, percentage, mean and standard deviation will be used as descriptive statistical methods in the evaluation of the data. Differences between the rates of categorical variables in independent groups are planned to be analyzed with Chi-Square tests. The t-test will be used to compare quantitative continuous data between two independent groups, and the changes in repeated measurements within the group will be analyzed with the dependent groups t-test.

Hypothesis(ies):

H1: Emotional Freedom Technique Applied to Mothers with Premature Babies in the Neonatal Intensive Care Unit reduces fatigue H2: Emotional Freedom Technique Applied to Mothers with Premature Babies in the Neonatal Intensive Care Unit Reduces Anxiety.

H3: Emotional Freedom Technique Applied to Mothers with Premature Babies in the Neonatal Intensive Care Unit increases mother-baby bonding.

DATA COLLECTION TOOLS AND FEATURES In data collection, the Introductory Information Form including socio-demographic characteristics, State-Trait Anxiety Scale (STAI I-II), Visual Similarity Scale for Fatigue (VAS-F) and Mother-Baby Attachment Scale (MIBS) will be used.

a. Introductory Information Form Information form prepared by the researchers in line with the literature; It consists of 32 questions containing information about socio-demographic characteristics such as age, gender, marital status, educational status, profession, and newborn and method satisfaction State-Trait Anxiety Inventory (STAI-II) The State-Trait Anxiety Inventory, consists of forty items and includes two separate scales, each with twenty items, which are completed by the patient themselves. its validity and reliability were tested. The Cronbach's alpha coefficient of the scale is 0.87. The inventory measures the state and trait anxiety levels of individuals and can be applied to healthy individuals aged 14 and above, as well as to patients who are mentally alert and able to understand and respond to questions. There is no time limit for the scale. The State-Trait Anxiety Inventory consists of four response categories: (1) Not at all, (2) A little, (3) Quite a bit, and (4) Completely for the state anxiety scale, and (1) Almost never, (2) Sometimes, (3) Often, and (4) Almost always for the trait anxiety scale. The higher the score obtained from the scale, the higher the individual's anxiety level. The total score obtained from the scale ranges from 20 to 80, where 20-39 indicates mild anxiety, 40-59 indicates moderate anxiety, 60-79 indicates high anxiety, and 80 indicates panic anxiety. The internal consistency and homogeneity coefficients, determined by alpha correlation, are reported to be between 0.94 and 0.96.

In this study, to determine the effect of the Emotional Freedom Technique (EFT) on the anxiety levels of mothers with premature babies in the neonatal intensive care unit, the State-Trait Anxiety Inventory will be applied three times: before the first EFT procedure within the first 24 hours after birth, immediately after the second EFT procedure one week following the first, and immediately after the second EFT procedure three weeks later.

Visual Similarity Scale for Fatigue (VAS-F) The scale consists of 18 items. Items 1, 2, 3, 4, 5, 11, 12, 13, 14, 15, 16, 17, and 18 are related to fatigue, while items 6, 7, 8, 9, and 10 are related to energy subscales. The Visual Similarity Scale for Fatigue consists of lines with a 10 cm long line between the most positive and the most negative expressions at each end. The items of the fatigue subscale move from the most positive to the most negative, while the energy subscale items go from the most negative to the most positive. A high score on the fatigue subscale and a low score on the energy subscale indicate a higher intensity of fatigue. Since the scoring range of the Visual Similarity Scale for Fatigue is not explicitly defined, it is considered to provide more sensitive measurements compared to scales with defined scoring ranges. Additionally, this scale is preferred due to its ease of use, brevity, and clarity.

Mother-Baby Attachment Scale (MIBS) This scale, designed to be used from the first day postpartum, allows the mother to describe her feelings toward her baby in a single word. It can be quickly and easily applie. The scale consists of 8 items and follows a 4-point Likert format. The items are answered with four options ranging from "(0) Very much" to "(3) Never." Items 1, 4, and 6 are positive emotional expressions and are scored 0, 1, 2, and 3, respectively. Items 2, 3, 5, 7, and 8 represent negative emotional expressions and are scored in reverse order: 3, 2, 1, and 0. The lowest score possible is 0, and the highest score is 24. As the score increases, the bonding is negatively affected. The inter-rater reliability of the scale is reported to be 0.71, and its internal consistency coefficient (Cronbach Alpha) is 0.66.

Data Collection Method The data collection tools will be applied to participants by the researcher. The data collection process will take approximately 60 minutes.

Steps of EFT Application in the Study

There are six steps involved in applying the EFT protocol. These steps have been prepared in accordance with the literature. The steps of the EFT application in this study are as follows:

Identifying the Problem and Rating the Emotion: Participants will be informed about the EFT protocol. The researcher will discuss the participants' feelings related to fatigue, anxiety, and bonding. The issue and the emotions it causes will be determined for the EFT protocol to be applied. To assess the intensity of the identified emotion, the participant will be asked to rate the emotion using the Subjective Units of Experience (SUE) scale while their eyes are closed in the "heart healing position".

Subjective Units of Experience Scale (SUE) The SUE scale, developed by Hartmann within the "Events Psychology" approach, is used to measure the energy flow in an individual's energy body. This scale is used at the beginning and end of the EFT session to determine the intensity of the participant's emotional state.

Scoring of the Scale The scale scores range from -10 to +10. "-10" represents the most intense pain, frustration, fear, stress, sadness, or discomfort imaginable.

"-1, 0, +1" represent a state of nothingness. There are no feelings, no inspiration, and no energy. Energy is needed here; there is no energy to take a step or begin something new.

"+10" corresponds to the highest levels of joy, happiness, or feeling great. Setup Statement Creation The setup statement involves clearly identifying the word or sentence that will help the participant recall the emotions evoked by the issue, and it is one of the most important factors affecting the success of the EFT technique . Examples of setup statements could include: "I'm worried about my baby's life," "I'm afraid something will happen to my baby," "I'm afraid my baby will become distant from me," "This process is exhausting me," "I haven't been able to rest since giving birth." The participant is encouraged to express these emotions and repeat them aloud during the session, in a way they can hear themselves. The setup statement must be clear, direct, and straightforward. The first half of the setup statement emphasizes exposure, while the second half contains the acceptance of the self. For example, in the second half, statements like "Even though I'm afraid something will happen to my baby, I love and accept myself," "Even though I have stress and anxiety about my baby's life, I choose to remain calm and forgive myself," and "Even though I'm exhausted, I choose to stay calm and rest" are used. The participant is then asked to repeat these sentences aloud in a way that they can hear themselves, acknowledging their feelings and self-acceptance.

Tapping After determining the emotional intensity based on the SUE scale, the tapping process begins under the guidance of the practitioner, following the sequence given in Figure 1. The tapping is done rhythmically on the EFT meridian points using the index and middle fingers, tapping 5-10 times on each point. The taps should not be too light to feel nothing, nor too hard to cause pain. During the tapping, the participant's eyes should be closed. The purpose of tapping is to remove blockages in the body's energy meridians and improve the flow of energy (Hartman, 2016). The first round will focus on negative EFT, while positive EFT will be done in the second and third rounds.

Affirmation After completing the negative round and the release round of the EFT protocol, the phase involves creating positive affirmation statements that will help the individual feel better and stronger emotionally in the face of their problem. Examples of positive affirmations include: "I accept my baby's premature birth," "My woman's body is in harmony/ready to bond with my baby," and "I choose to be calm in the face of my worries." These positive affirmation sentences are created with the woman's chosen words.

Reevaluation In the final stage of the EFT protocol, the participant will move to the "heart healing point," take three deep breaths, and then reassess themselves on the SUE scale in comparison to the beginning. Affirmations will continue until emotions reach a neutral "0" point.

Implementation of the Research The EFT sessions will be conducted by the researcher who holds an E-government certified EFT Expertise certificate.

The study consists of two groups: an intervention group and a control group. Mothers with premature babies in the neonatal intensive care unit will be randomly selected for both the intervention and control groups.

Limitations of the Study A limitation of this study is the inclusion of mothers with premature babies only from two centers: Bezmialem Vakif University Center and Dragos Hospitals. The results obtained from the study can be generalized to this specific group.

Steps for the Intervention Group:

Pre-Intervention:

* Participants in the intervention group will be informed about EFT, and after explaining the aim and method of the study, their consent will be obtained using the Volunteer Consent Form.
* They will complete the State-Trait Anxiety Inventory (STAI-I-II), and those who score 40 or higher will be included in the study.
* Afterward, information will be provided about EFT, including how the procedure will be performed and how tapping will be done. Following a discussion planned to last approximately 20 minutes, the EFT session will begin.
* Prior to the intervention, women will be asked to fill out the Descriptive Information Form, State-Trait Anxiety Inventory , Visual Similarity Scale for Fatigue , and Mother-Infant Bonding Scale forms.

  1. EFT Procedure Sequence:
* The first meeting will be conducted within the first 24 hours after the admission of mothers who meet the inclusion criteria for our study in the NICU.
* The mother will be ensured to be in an environment where she feels alone, relaxed, and safe.

EFT Session: The EFT session will be conducted mutually with the practitioner. The average duration of the session is planned to be 40-45 minutes.

After the session, affirmation sentences will be provided for the mother to repeat with tapping for 3 days. Every day, the mother will be asked whether she has repeated the affirmation sentences. This will be monitored through a prepared chart (Appendix 6).

2. EFT Procedure Sequence: One week after the first EFT session, the second session will be conducted for the intervention group. This session is planned to last approximately 45 minutes.

Immediately after the first EFT session, the State-Trait Anxiety Inventory (STAI-I-II), Visual Similarity Scale for Fatigue (VAS-F), and Mother-Infant Bonding Scale (MIBS) forms will be administered.

3. EFT Procedure Sequence: Three weeks after the second EFT session, the techniques included in the EFT will be applied to the women in the intervention group for an average of 40-45 minutes.

Immediately after the third EFT session, the State-Trait Anxiety Inventory (STAI I-II), Visual Similarity Scale for Fatigue (VAS-F), and Mother-Infant Bonding Scale (MIBS) will be administered, along with questions about the satisfaction with the application.

Control Group Application Steps Control Group 1st Meeting (Pre-test): The mothers in the control group, who have premature babies in the neonatal intensive care unit, will be informed about the study. After explaining the purpose and method of the study, their consent will be obtained through the Volunteer Consent Form.

The women will complete the forms, and those with a score of 40 or above will be included in the study.

The women in the control group will be asked to complete the Descriptive Information Form, State-Trait Anxiety Inventory (STAI I-II), Visual Similarity Scale for Fatigue (VAS-F), and Mother-Infant Bonding Scale (MIBS) forms.

No intervention will be provided for the mothers in the control group, but the institution's neonatal intensive care services will be available to them.

Control Group 2nd Meeting: One week after the first meeting, the State-Trait Anxiety Inventory (STAI I-II), Visual Similarity Scale for Fatigue (VAS-F), and Mother-Infant Bonding Scale (MIBS) forms will be administered again.

Control Group 3rd Meeting: Three weeks after the first meeting, the State-Trait Anxiety Inventory (STAI I-II), Visual Similarity Scale for Fatigue (VAS-F), and Mother-Infant Bonding Scale (MIBS) forms will be administered again.

DATA ANALYSIS METHOD The data obtained in the research will be analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. Descriptive statistical methods such as frequency, percentage, mean, and standard deviation will be used to evaluate the data. Differences in the proportions of categorical variables between independent groups are planned to be analyzed using Chi-Square tests. The t-test will be used to compare quantitative continuous data between two independent groups, and the changes in repeated measurements within the group will be analyzed using the dependent groups t-test. The Kolmogorov-Smirnov Test will be used to determine whether the research data is normally distributed. If p > 0.05 in the Kolmogorov-Smirnov Test, the distribution will be considered normal. However, if p < 0.05, the distribution will be considered non-normal, and the values of Skewness and Kurtosis will be examined. If the Skewness and Kurtosis values are between +2 and -2, the variable will be accepted as normally distributed. The homogeneity of descriptive characteristics between groups will be tested using the chi-square analysis. To evaluate the difference between the means of two independent groups, if the data is normally distributed, the t-test will be used; if the data is not normally distributed, the Mann-Whitney U test will be used. For changes in measurements within the group, if the data is normally distributed, the repeated measures ANOVA will be used; if the data is not normally distributed, the Friedman test will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Those who can read and write and who can speak and understand Turkish,
* Those whose STAI-I (status) score range is 40 and above
* Mothers whose babies were born prematurely
* Mothers whose babies are in NICU,
* Mothers who agreed to participate in the study.

Exclusion Criteria:

* Mothers of premature newborns who cannot be fed with breast milk,
* Mothers who were discharged during the study sessions and did not agree to continue working,
* The mother has any cognitive or hearing-related problems,
* The mother has a psychiatrically diagnosed disease (Schizophrenia, bipolar disorder, depression).
* Having epilepsy (since it is contraindicated for EFT applications)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — puerperıum
Enrollment: 64 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Fatigue, Anxiety, and Mother-Baby Bonding and Effect of the Emotional Freedom | 2 year
  1. Visual Similarity Scale for Fatigue (VSSF): This is a visual analog scale designed to assess an individual's subjective level of fatigue. Participants are presented with a straight line anchored by the descriptors "not at all fatigued" (0 points) on one end and "extremely fatigued" (10 points) on the other. Participants are asked to mark the point on the line that best represents their current fatigue level. Scores range from a minimum of 0 to a maximum of 10. Higher scores indicate a higher level of perceived fatigue. This scale is widely used in clinical settings due to its simplicity and efficiency.
Fatigue, Anxiety, and Mother-Baby Bonding and Effect of the Emotional Freedom | 2 year
  2.State-Trait Anxiety Inventory (STAI-II) The State-Trait Anxiety Inventory (STAI-II) consists of two subscales that measure state and trait anxiety, each using a four-point Likert-type response format. In the State Anxiety Scale, the response options are: (1) Not at all, (2) Somewhat, (3) Moderately so, and (4) Very much so. In the Trait Anxiety Scale, the options are: (1) Almost never, (2) Sometimes, (3) Often, and (4) Almost always. Higher scores on the inventory indicate a higher level of anxiety. The total score obtained from the scale ranges between 20 and 80. Scores between 20 and 39 indicate mild anxiety, scores between 40 and 59 indicate moderate anxiety, scores between 60 and 79 indicate high anxiety, and a score of 80 indicates a panic-level anxiety.
Fatigue, Anxiety, and Mother-Baby Bonding and Effect of the Emotional Freedom | 2 year
  3.Mother-Infant Bonding Scale (MIBS) The Mother-Infant Bonding Scale is designed to be used from the very first day after birth and allows the mother to describe her feelings toward her baby in a single word. The scale consists of 8 items and is structured as a 4-point Likert-type scale. Each item is rated using four response options ranging from (0) Very much to (3) Never. Items 1, 4, and 6 reflect positive emotions and are scored as 0, 1, 2, 3 respectively. Items 2, 3, 5, 7, and 8 reflect negative emotions and are reverse scored as 3, 2, 1, 0. The total score ranges from 0 to 24, with higher scores indicating more negative effects on bonding between the mother and the baby.

CONTACTS AND LOCATIONS:
Overall Officials: HANDAN ÖZCAN, Associate Professor, Study Director — HAMİDİYE HEALTH SCİENCE UNIVERSTY

IPD SHARING:
Plan to Share IPD: No